CLINICAL TRIAL: NCT01202292
Title: Group Motivational Intervention in Overweight/Obese Patients in Primary Prevention of Cardiovascular Disease in the Primary Healthcare Area.
Brief Title: Group Motivational Intervention in Overweight/Obese Patients.
Acronym: IMOAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Juan José Rodriguez Cristóbal, ABS FLORIDA SUR
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PI 070087
Record Dates: First submitted 2010-05-31; First posted 2010-09-15 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; motivational intervention
MeSH Terms: conditions — Overweight; Obesity | interventions — Psychotherapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling)

INTERVENTIONS:
Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) — Group motivational intervention consist in expert psychologist 32 monthly sessions (group intervention) on top of the diet plus exercise
  Other Names: Control group receives the usual follow up: diet, exercise

SUMMARY:
The overall goal of IMOAP study is to assess whether the efficacy of the healthcare professionals' usual practices, together with a motivational group intervention (delivered by a nurse trained by an expert psychologist), is more effective than an isolated traditional intervention on weight loss and its maintenance in overweight and obese patients. Furthermore, the study will evaluate whether this result has a positive impact on quality of life, changes in eating habits, and a reduction in the associated cardiovascular risk factors and overall cardiovascular risk.

DETAILED DESCRIPTION:
The global mortality caused by cardiovascular disease increases with weight. The Framingham study showed that obesity is a cardiovascular risk factor independent of other risks such as type 2 diabetes mellitus, dyslipidemia and smoking. Moreover, the main problem in the management of weight-loss is its maintenance, if it is achieved. We have designed a study in two geographically separated groups, one of which would receive the group motivational intervention, and the other one would receive the usual follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight (BMI>25) and obese (BMI>30) patients of both sexes, registered in the medical history (MH) or newly diagnosed.
2. Aged between 30 and 70 years
3. Agreement to participate in the study

Exclusion Criteria:

1. Patients with severe clinical pathology (bedridden, dementia, advanced neoplasia, etc.)
2. Patients with secondary obesity (hypothyroidism, Cushing's disease, etc)
3. Patients with severe sensorial disorders capable of interfering with the motivational intervention (severe, uncorrected deafness, severe visual deficit, etc).
4. Patients with serious psychiatric disorders

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Determine whether a group motivational intervention, is more efficient than the latter in the treatment of overweight and obesity, for initial weight loss and essentially to achieve sustained normalisation of the weight achieved. | 26 months

SECONDARY OUTCOMES:
Observe whether this intervention is more effective for reducing cardiovascular risk factors associated to overweight and obesity, and in the overall cardiovascular risk in these patients. | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Roodriguez-Cristóbal, Dr, Principal Investigator — Catalan Institute of Health
Locations (1):
- ABS Florida Sud, L'Hospitalet Del Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Rodriguez Cristobal JJ, Panisello Royo JM, Alonso-Villaverde Grote C, Perez Santos JM, Munoz Lloret A, Rodriguez Cortes F, Trave Mercade P, Benavides Marquez F, Marti de la Morena P, Gonzalez Burgillos MJ, Delclos Baulies M, Bleda Fernandez D, Quillama Torres E; IMOAP Group. Group motivational intervention in overweight/obese patients in primary prevention of cardiovascular disease in the primary healthcare area. BMC Fam Pract. 2010 Mar 18;11:23. doi: 10.1186/1471-2296-11-23. PMID 20298557